CLINICAL TRIAL: NCT03813186
Title: A Phase 1b Study to Evaluate the Effect of Food on Pharmacokinetics of ASTX727 (Cedazuridine and Decitabine) in Subjects With Myelodysplastic Syndromes or Acute Myeloid Leukemia
Brief Title: Effect of Food on Blood Levels of ASTX727
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ASTX727-04
Record Dates: First submitted 2019-01-11; First posted 2019-01-23 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Acute Myeloid Leukemia
Keywords: MDS; CMML; ASTX727; decitabine; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; cedazuridine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASTX727 + Day 2 Food (Experimental): Subjects will receive ASTX727 on Days 1-5 of Cycle 1 and a high-calorie, high-fat breakfast meal of 800-1000 calories pre-dose on Day 2 of Cycle 1.
  Interventions: Drug: ASTX727 + Day 2 Food
- ASTX727 + Day 4 Food (Experimental): Subjects will receive ASTX727 on Days 1-5 of Cycle 1 and a high-calorie, high-fat breakfast meal of 800-1000 calories pre-dose on Day 4 of Cycle 1.
  Interventions: Drug: ASTX727 + Day 4 Food

INTERVENTIONS:
Drug: ASTX727 + Day 2 Food — ASTX727 is an oral drug product composed of a fixed-dose combination of cedazuridine (E7727), a CDA inhibitor, and decitabine. Food is a high-calorie, high-fat breakfast meal of 800-1000 calories given on Day 2.
  Other Names: cedazuridine + decitabine + food on Day 2
  Arms: ASTX727 + Day 2 Food
Drug: ASTX727 + Day 4 Food — ASTX727 is an oral drug product composed of a fixed-dose combination of cedazuridine (E7727), a CDA inhibitor, and decitabine. Food is a high-calorie, high-fat breakfast meal of 800-1000 calories given on Day 4.
  Other Names: cedazuridine + decitabine + food on Day 4
  Arms: ASTX727 + Day 4 Food

SUMMARY:
This study is designed to examine blood levels of ASTX727, a fixed-dose combination tablet containing the combination of cedazuridine (100 mg) and decitabine (35 mg), when given under fed versus fasted conditions to participants with myelodysplastic syndromes (MDS), including refractory anemia with excess blasts in transformation or chronic myelomonocytic leukemia (CMML), or acute myeloid leukemia (AML). This study will also assess the safety of ASTX727.

DETAILED DESCRIPTION:
This is a Phase 1b, multicenter, open-label, randomized, two-sequence, crossover study of ASTX727 in participants with MDS, including refractory anemia with excess blasts in transformation or CMML, and AML. Participants will continue to be enrolled until evaluable data is collected from 12 participants. It is expected that approximately 18 participants will be enrolled in total.

This study will be conducted in 28-day cycles. All participants will take part in Cycle 1 and may continue into Cycles ≥2 at the investigator's discretion. Participants will receive one tablet of ASTX727 containing 100 mg cedazuridine and 35 mg decitabine once daily for 5 days in 28-day cycles starting from Cycle 1 Day 1.

Participants will be randomized in a 1:1 ratio to receive high-calorie, high-fat breakfast meal pre-dose on either Day 2 or Day 4 of Cycle 1. Blood will be drawn at specified time points in Cycle 1 on Days 2 through 5 to assess the effect of food on the PK of cedazuridine and decitabine.

After completion of the first treatment cycle, participants may continue to receive treatment with ASTX727 at the investigator's discretion for subsequent cycles (Days 1 through 5 of 28-day cycles), until disease progression, unacceptable toxicity, investigator decision to discontinue treatment, or the participant decides to discontinue treatment or withdraw from the study. In Cycles ≥2, participants will fast for 2 hours before and 2 hours after taking the ASTX727 tablet on all dosing days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, including the ability to completely consume the breakfast meal in 20 minutes, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure.
2. Men or women ≥18 years with either:

   1. MDS, including all French-American-British subtypes (refractory anemia, refractory anemia with ringed sideroblasts, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, CMML), and subjects with MDS IPSS int-1, -2, or high-risk MDS.
   2. AML, as diagnosed according to the 2016 WHO guidelines on acute leukemia, of any subtype except M3 (Acute Promyelocytic Leukemia), who are not candidates for intensive chemotherapy
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Adequate organ function defined as follows:

   1. Hepatic: Total or direct bilirubin ≤2 × upper limit of normal (ULN); aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) ≤5 × ULN.
   2. Renal: serum creatinine ≤1.5 × ULN or if serum creatinine is elevated; calculated creatinine clearance or glomerular filtration rate ≥50 mL/min.
5. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.
6. Subjects and their partners with reproductive potential must agree to use 2 highly effective contraceptive measures during the study and must agree not to become pregnant or father a child for 3 months after the last dose of study treatment.

Exclusion Criteria:

1. Known or suspected hypersensitivity to decitabine, azacitidine, or cedazuridine.
2. Treated with any investigational drug or therapy within 2 weeks of study treatment, or 5 half-lives, whichever is longer, before the protocol-defined first dose of study treatment, or ongoing clinically significant adverse events (AEs) from previous treatment with investigational drug or therapy.
3. Poor medical risk because of other conditions such as uncontrolled systemic diseases or active uncontrolled infections.
4. Life-threatening illness, medical condition or organ system dysfunction, or other reasons including laboratory abnormalities, which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of decitabine + cedazuridine or compromise the integrity of the study outcomes.
5. Prior gastric surgery for ulcer disease, weight loss, etc., that would impair normal motility or absorption.
6. Second malignancy currently requiring active chemotherapy. To clarify, patients with breast or prostate cancer stable on or responding to endocrine therapy, are eligible.
7. Known history of human immunodeficiency virus or if known seropositive for hepatitis C virus or hepatitis B virus.
8. Active uncontrolled gastric or duodenal ulcer.
9. Subjects with Acute Promyelocytic Leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
AUC0-t (area under the concentration-time curve from time 0 to t hours). | 6 months
  Area under the concentration-time curve from time 0 to t hours.
AUC0-8 (area under the concentration-time curve from time 0 to 8 hours). | 6 months
  Area under the concentration-time curve from time 0 to 8 hours.
AUC0-24 (area under the concentration-time curve from time 0 to 24 hours). | 6 months
  Area under the concentration-time curve from time 0 to 24 hours
AUC0-inf (area under the concentration-time curve from time 0 to infinity). | 6 months
  Area under the concentration-time curve from time 0 to infinity.
Cmax (maximum plasma concentration). | 6 months
  Maximum plasma concentration.

SECONDARY OUTCOMES:
hemoglobin level | 6 months
  Assessed in g/dL
platelet count | 6 months
  Assessed as 10^9/L
white blood cell count | 6 months
  Assessed as fraction of 1
neutrophils | 6 months
  Assessed as percent
Subject-reported and investigator-observed incidence and severity of adverse events. | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Roswell Park, Buffalo, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Vanderbilt, Nashville, Tennessee
  - Mays Cancer Center UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072